CLINICAL TRIAL: NCT06951776
Title: Chronotherapeutic Optimization of Teriparatide Administration in Postmenopausal Osteoporosis: A Randomized Controlled Exploratory Study
Brief Title: Chronotherapeutic Optimization of Teriparatide Administration in Postmenopausal Osteoporosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20250309
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Circadian Rhythm Disorders; Osteoporosis
Keywords: Teriparatide, osteoporosis, Chronotherapy
MeSH Terms: conditions — Chronobiology Disorders; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Twenty-eight participants (age 60-70 years, lumbar spine T-score ≤-3.0) will undergo 1:1 randomization to receive 20 µg/day teriparatide subcutaneously at either 08:00 or 20:00 for 12 weeks. Standardized supplementation with calcium (1,000-1,500 mg/day) and cholecalciferol (800-1,200 IU/day) will be maintained. Primary endpoints are between-group differences in serum CTX and P1NP profiles, quantified at baseline, 4-week interim, and 12-week endpoint. The secondary outcomes will assess safety during the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning (8:00) administration group of teriparatide (Experimental): A total of 14 subjects will be included. Teriparatide injection (20 µg, subcutaneous injection, once daily) will be administered in the morning (around 8:00 a.m.) every day for 12 weeks
  Interventions: Behavioral: Morning administration group of teriparatide
- Evening (20:00) administration group of teriparatide (Experimental): A total of 14 subjects will be included. Teriparatide injection (20 µg, subcutaneous injection, once daily) will be administered in the evening (around 20:00 p.m.) every day for 12 weeks
  Interventions: Behavioral: Evening administration group of teriparatide

INTERVENTIONS:
Behavioral: Morning administration group of teriparatide — Eligible participants will be randomly assigned (1:1) to either subcutaneous injection of 20 μg teriparatide at 08:00 a.m. in the morning (Group A) and subcutaneous injection of 20 μg teriparatide at 20:00 p.m. in the evening (Group B).
  Arms: Morning (8:00) administration group of teriparatide
Behavioral: Evening administration group of teriparatide — Eligible participants will be randomly assigned (1:1) to either subcutaneous injection of 20 μg teriparatide at 08:00 a.m. in the morning (Group A) and subcutaneous injection of 20 μg teriparatide at 20:00 p.m. in the evening (Group B).
  Arms: Evening (20:00) administration group of teriparatide

SUMMARY:
This is a randomized, controlled, and exploratory study designed to evaluate the chronotherapeutic effects of teriparatide administration in postmenopausal osteoporosis. Twenty-eight participants (age 60-70 years, lumbar spine T-score ≤-3.0) will undergo 1:1 randomization to receive 20 µg/day teriparatide subcutaneously at either 08:00 or 20:00 for 12 weeks. Standardized supplementation with calcium (1,000-1,500 mg/day) and cholecalciferol (800-1,200 IU/day) will be maintained. Primary endpoints are between-group differences in serum CTX and P1NP profiles, quantified at baseline, 4-week interim, and 12-week endpoint. The secondary outcomes will assess safety during the trial.

DETAILED DESCRIPTION:
This is a randomized, controlled, and exploratory study designed to evaluate the chronotherapeutic effects of teriparatide administration in postmenopausal osteoporosis. The trial protocol was approved by the Peking University Third Hospital Medical Science Research Ethics Committee. This trial intends to enroll postmenopausal osteoporosis patients admitted to the Department of Orthopedics of Peking University Third Hospital. Subjects who meet the inclusion and exclusion criteria can be enrolled in this trial after signing the informed consent form. Each trial group plans to enroll 14 subjects, with a total of 28 subjects. Eligible participants will be randomly assigned (1:1) to either subcutaneous injection of 20 μg teriparatide at 08:00 a.m in the morning (Group A) and subcutaneous injection of 20 μg teriparatide at 20:00 p.m in the evening(Group B). The specific time of drug administration for each patient every day needs to be recorded in the diary card. All subjects will be given calcium (1000-1500 mg/day) and vitamin D (800-1200 IU/day) simultaneously during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60-70 years (inclusive).
2. Naturally postmenopausal women with≥5 years since last menses.
3. DXA-measured BMD T-score≤-3.0 at lumbar spine (L1-L4) and/or total hip at screening.
4. The concentration of 25-hydroxyvitamin D (25-OH)D is ≥20 ng/ml. If the subject meets all other inclusion and exclusion criteria, it is allowed to retest the 25-OHD concentration after administering vitamin D to the subject.
5. Normal-range serum parameters:

Intact PTH: 15-65 pg/mL Total calcium: 2.20-2.70 mmol/L.

Exclusion Criteria:

1. Subjects with bone metabolic diseases besides osteoporosis:

   1. Other metabolic bone diseases, such as osteomalacia, osteogenesis imperfecta, Paget's disease；
   2. Cushing's syndrome;
   3. Hyperprolactinemia;
2. Use of medications that affect bone metabolism before screening:

   Use of intravenous bisphosphonates, fluoride, or strontium within 2 years; Use of teriparatide or denosumab for osteoporosis within 6 months; Oral bisphosphonates for osteoporosis with the last dose within 1 year (if used within 1 year but with a cumulative use of ≤1 month, the subject is eligible); Continuous use of calcitonin for more than 3 months with the last dose within 1 year.
3. History of malignancy within 5 years, or bone metastasis, except for tumors that are expected to be cured after treatment (such as completely resected in situ basal cell or squamous cell carcinoma of the skin, cervical cancer, or breast ductal carcinoma, etc.).
4. Hypocalcemia and hypercalcemia.
5. Elevated alkaline phosphatase of unknown cause.
6. History of fractures.
7. Uncontrolled comorbidities, including heart failure with New York Heart Association (NYHA) functional class III or above, glycated hemoglobin >8.5%, and severe arrhythmias.
8. Allergy to teriparatide.
9. Currently participating in another drug clinical trial.
10. Subjects deemed unsuitable for enrollment in this study by the investigator.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of CTX from baseline after administration | Within 12 weeks
  Compare the morning and evening dosing groups regarding the changes in serum CTX from baseline after 4 and 12 weeks of subcutaneous injection of teriparatide.
Change of P1NP from baseline after administration | Within 12 weeks
  Compare the morning and evening dosing groups regarding the changes in serum P1NP from baseline after 4 and 12 weeks of subcutaneous injection of teriparatide.
Change of PTH from baseline after administration | Within 12 weeks
  Compare the morning and evening dosing groups regarding the changes in serum PTH from baseline after 4 and 12 weeks of subcutaneous injection of teriparatide.

SECONDARY OUTCOMES:
Safety Evaluation | Within 12 weeks
  All adverse drug reactions that occurred during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, Dr, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Tao L, Liu D, Yan X, Li H, Song C. Timing optimization of teriparatide dosing for postmenopausal osteoporosis: a randomized controlled trial. J Orthop Surg Res. 2025 Jul 17;20(1):669. doi: 10.1186/s13018-025-06083-6. PMID 40676595